CLINICAL TRIAL: NCT07349940
Title: Early Detection of Skin Tumors Using a Telemedicine Tool in Primary Care
Acronym: MEL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: University Hospital Kralovske Vinohrady (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UZIS 2025/6
Record Dates: First submitted 2025-11-18; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Skin Cancer Prevention; Melanoma In Situ; Skin Lesions; Skin Cancer; Mole (Dermatology)
Keywords: skin cancer; melanoma; telemedicine tool; skin tumors
MeSH Terms: conditions — Skin Neoplasms; Nevus; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with suspected skin lession (Experimental): Pilot screening will be conducted in general practitioners' offices, where physicians will be trained to examine skin lesions using magnifying devices (dermatoscopes) and advanced telemedicine software, enabling faster diagnostics of suspicious findings. Patients with high-risk lesions will be referred to specialized dermatology centers.
  Interventions: Diagnostic Test: Intervention with telemedicine tool

INTERVENTIONS:
Diagnostic Test: Intervention with telemedicine tool — The diagnostic management of enrolled patients will be guided by standardized procedures carried out in general practitioners' offices. Physicians will be trained to identify suspicious skin lesions, capture high-resolution images using dermatoscopes, and transfer the data into advanced telemedicine software. The platform, supported by AI-driven algorithms, enables precise risk stratification of lesions and facilitates remote consultation with collaborating dermatologists.
  Patients with high-risk lesions will be referred to specialized dermatology centers for further examination and intervention. In cases where excision of a lesion is performed, histopathological assessment will be conducted, and results will be systematically recorded within the dedicated telemedicine platform, ensuring secure and efficient information exchange between dermatologists and general practitioners.

SUMMARY:
The project is a national, prospective, multicenter, single-arm interventional pilot of screening skin tumors in the Czech Republic.

The primary aim of the project is to methodically prepare, implement and evaluate a pilot project that will verify the suitability of the proposed procedure of early detection of skin tumors by using a telemedicine tools and setting up and testing new methods and implementation into the system of social health care.

DETAILED DESCRIPTION:
The project is a national, prospective, multicenter, single-arm interventional pilot project for skin tumors screening involving 18 general practitioners and 6 dermatology centers in the Czech Republic.

The main objective of the project is the early detection of skin tumors by general practitioners, increasing the efficiency of healthcare, and methodically preparing, implementing, and evaluating the pilot project. The project aims to verify the suitability of the proposed early detection procedure for skin tumors, as well as to establish and test new methods and integrate them into the healthcare system.

As part of the project, the procedure will be tested on a sample of approximately 1,440 individuals, which may help validate the use of telemedicine tools in healthcare. A methodology for the use of telemedicine tools will be developed, along with a framework for collaboration between general practitioners and affiliated dermatologists. Systemic changes will be proposed to enhance the efficiency of the screening process.

The project is supported by the European Social Fund (Operational Programme Employment Plus) and the state budget of the Czech Republic. It is registered with the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.02.02/00/22_005/0002008.

ELIGIBILITY:
Inclusion Criteria:

* at least 1 suspected lession
* phototype I or phototype II

Exclusion Criteria:

* skin lession examination by dermatologist in last 12 months
* unsigned consent to participate in the project and consent to the processing of personal data

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Potential malignancies | From enrollment to the end of examination - baseline.
  Proportion of individuals with a potential presence of malignancy (detected through the telemedicine tool).
Confirmed malignancies | From enrollment to the end of diagnosis at 3 months.
  Proportion of individuals with confirmed potential malignancy by a dermatologist.
Confirmed malignancies by histology | From enrollment to the end of diagnosis at 6 months.
  Proportion of individuals in whom the diagnosis of malignancy was confirmed histologically.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Arenberger, prof., Study Director — Hospital university Kralovske Vinohrady
Locations (5):
- Czechia (5):
  - St. Anne's University Hospital Brno, Brno
  - Olomouc University Hospital, Olomouc
  - University Hospital Pilsen, Pilsen
  - Bulovka University Hospital, Prague
  - University hospital Kralovske Vinohrady, Prague

IPD SHARING:
Plan to Share IPD: No